CLINICAL TRIAL: NCT06556355
Title: Impact of Preoperative Radiation Dose to the Cervical Esophagus on Anastomotic Leak in Esophageal Squamous Cell Carcinoma Patients After Neoadjuvant Chemoradiation and McKeown Esophagectomy: A Retrospective Analysis
Brief Title: Anastomotic Leaks in Esophageal Squamous Cell Carcinoma Patients After Trimodal Therapy
Status: Completed | Type: Observational
Sponsor: Qiaoqiao Li (Other)
Collaborators: Chinese Institute of Food Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Qiaoqiao Li, Chief Medical Officer, Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Other Study IDs: 202210172055000282645
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Anastomotic Leak Esophagus
Keywords: esophageal cancer; anastomotic leak; neoadjuvant chemoradiation; radiation dose; esophagectomy; outcomes
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall patients: Consecutive patients with locally advanced thoracic ESCC who underwent nCRT and surgery at our center between 1 January 2015 and 31 December 2020.
  Interventions: Other: neoadjuvant chemoradiation and McKeown esophagectomy

INTERVENTIONS:
Other: neoadjuvant chemoradiation and McKeown esophagectomy — Treatment protocol:
  1. All patients were irradiated a total prescribed dose of 40-50.4 Gy in 20-28 fractions by a 6-8 MV photons linear accelerator with the intensity-modulated radiotherapy or volumetric modulated arc therapy technique.
  2. Concurrent chemotherapy was cisplatin-based.
  3. McKeown esophagectomy (three incision) consisted of thoracic esophageal mobilization with lymphadenectomy, abdominal exploration and stomach mobilization with lymphadenectomy, and subsequently left cervical incision for anastomosis. The lymphadenectomy was total two-field (thoracic + abdomen).

SUMMARY:
To investigate the clinical factors and preoperative treatment to the future anastomotic location of cervical esophagus that were correlated with anastomotic leaks in esophageal squamous cell carcinoma patients undergoing neoadjuvant chemoradiation and McKeown esophagectomy and to explore the prognosis of anastomotic leak.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the clinical factors and preoperative treatment to the future anastomotic location of cervical esophagus that were correlated with anastomotic leaks in esophageal squamous cell carcinoma patients undergoing neoadjuvant chemoradiation and McKeown esophagectomy and to explore the postoperative complications, mortality, and long-term survival of different types of anastomotic leak.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed ESCC;
* clinically staged as T3-4aN0M0 or T1-4aN+M0 by the eighth edition of the American Joint Committee on Cancer and treated with nCRT followed by McKeown esophagectomy24;
* aged 18-75 years;
* Eastern Cooperative Oncology Group performance status score ≤ 2.

Exclusion Criteria:

* cervical esophageal cancer;
* previously treated with chest radiotherapy, esophageal, or gastric surgery;
* insufficient clinical data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with locally advanced thoracic ESCC who underwent nCRT and surgery at our center between 1 January 2015 and 31 December 2020 were retrospectively identified and analyzed.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
anastomotic leak rate | Up to 1 month
  According to the consensus on standardization of data collection for complications associated with esophagectomy by the Esophagectomy Complications Consensus Group (ECCG), anastomotic leak was defined as a full-thickness gastrointestinal defect involving the esophagus, anastomosis, staple line or conduit, which was diagnosed as extravasation of water-soluble contrast during a swallow study, postoperative esophageal barium X-ray or CT scan, visualization of anastomotic dehiscence or leak during endoscopy, or salivary fluid in the cervical region.

SECONDARY OUTCOMES:
Overall survival | From date of pathological diagnosis until the date of death from any cause or censoring, assessed up to 36 months
  Overall survival (OS) was defined as the duration from the date of pathological diagnosis to the date of death or censoring.

OTHER OUTCOMES:
Pathologic complete response | Up to 1 month
  Pathologic complete response (pCR) was defined as no evidence of residual tumor cells in the primary tumors and resected lymph nodes of the operative specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Qiaoqiao Li, Study Chair — Sun Yat-sen University Cancer Center, Guangzhou, China; Chen Yang, Principal Investigator — Sun Yat-sen University Cancer Center, Guangzhou, China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The research data are stored in an institutional repository and will be shared on reasonable request from the corresponding author.
Supporting Information: CSR